CLINICAL TRIAL: NCT01258101
Title: Randomized, Multicenter Study to Compare the Efficacy of Pegylated Interferon Alfa (PEG-IFN) in Combination With Two Different Doses of Ribavirin in Patients With Chronic Hepatitis C and Subtype 2/3
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a) Plus Ribavirin in Patients With Chronic Hepatitis C (CHC), Genotype 2 or 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17087
Record Dates: First submitted 2010-11-29; First posted 2010-12-10 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (4):
- Peginterferon/Ribavirin 800 mg (24 Weeks) (Experimental): Participants received peginterferon alfa-2a (PEG-IFNα-2a) 180 mcg once weekly + Ribavirin 800 mg daily for 24 weeks (W).
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin
- Peginterferon/Ribavirin 400 mg (24 Weeks) (Experimental): Participants received PEG-IFNα-2a 180 mcg once weekly + Ribavirin 400 mg daily for 24 W.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin
- Peginterferon/Ribavirin 800 mg (16 Weeks) (Experimental): Participants received PEG-IFNα-2a 180 mcg once weekly + Ribavirin 800 mg daily for 16 W.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin
- Peginterferon/Ribavirin 400 mg (16 Weeks) (Experimental): Participants received PEG-IFNα-2a 180 mcg once weekly + Ribavirin 400 mg daily for 16 W.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 24 weeks
  Arms: Peginterferon/Ribavirin 400 mg (24 Weeks); Peginterferon/Ribavirin 800 mg (24 Weeks)
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 16 weeks
  Arms: Peginterferon/Ribavirin 400 mg (16 Weeks); Peginterferon/Ribavirin 800 mg (16 Weeks)
Drug: ribavirin — 800 mg orally daily
  Arms: Peginterferon/Ribavirin 800 mg (16 Weeks); Peginterferon/Ribavirin 800 mg (24 Weeks)
Drug: ribavirin — 400 mg orally daily
  Arms: Peginterferon/Ribavirin 400 mg (16 Weeks); Peginterferon/Ribavirin 400 mg (24 Weeks)

SUMMARY:
This randomized, parallel arm study will evaluate the efficacy and safety of Pegasys (peginterferon alfa-2a) in combination with 2 different doses of ribavirin in patients with chronic hepatitis C, genotype 2 or 3. Patients will be randomized to 4 treatment groups receiving Pegasys (180 mcg subcutaneously weekly) for either 16 or 24 weeks with one of two doses of ribavirin (400 mg or 800 mg orally daily). The anticipated time on study treatment is 16 or 24 weeks with a 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* Chronic hepatitis C, genotype 2 or 3
* Positive HCV RNA level in serum at screening (COBAS AMPLICOR MONITOR HCV test)
* Abdominal sonography within 3 months prior to study start

Exclusion Criteria:

* Previous interferon and/or pegylated interferon and ribavirin therapy
* Liver cirrhosis, class B or C (Child-Pugh)
* Systemic anti-neoplastic or immunomodulatory treatment <=6 months before study drug
* History or evidence of medical condition associated with chronic liver disease other than chronic hepatitis C
* Decompensated liver disease
* Positive for HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2003-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- Austria (11):
  - Gratwein
  - Graz
  - Innsbruck
  - Linz
  - Oberndorf
  - Ried-innkreis
  - Salzburg
  - Vienna
  - Villach
  - Wels
  - Wiener Neustadt

REFERENCES:
- [Derived] Maieron A, Metz-Gercek S, Scherzer TM, Laferl H, Fischer G, Bischof M, Gschwantler M, Ferenci P. Shortening of treatment duration in patients with chronic hepatitis C genotype 2 and 3 - impact of ribavirin dose - a randomized multicentre trial. BMC Res Notes. 2011 Jun 29;4:220. doi: 10.1186/1756-0500-4-220. PMID 21714878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 395 participants were recruited at 20 centres in Austria in the study conducted from 20 May 2003 to 10 July 2008.
Pre-assignment Details: Of the 395 participants, 380 were randomized to treatment groups. A total of 15 participants were screening failures.
Groups:
- Peginterferon/Ribavirin 800 mg (24 Weeks): Eligible participants were administered peginterferon alfa-2a (PEG-IFNα-2a) 180 microgram (mcg) subcutaneously (SC) once weekly + Ribavirin 800 milligram (mg) orally daily for 24 weeks (W). The untreated Follow-up was for 24 W.
- Peginterferon/Ribavirin 400 mg (24 Weeks): Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 400 mg orally daily for 24 W. The untreated Follow-up was for 24 W.
- Peginterferon/Ribavirin 800 mg (16 Weeks): Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 800 mg orally daily for 16 W. The untreated Follow-up was for 24 W.
- Peginterferon/Ribavirin 400 mg (16 Weeks): Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 400 mg orally daily for 16 W. The untreated Follow-up was for 24 W.
Period: Overall Study
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Started | 151 | 144 | 33 | 52
Safety Analysis Population | 144 | 141 | 30 | 48
Standard Analysis Population | 115 | 110 | 21 | 26
Completed | 118 | 110 | 22 | 27
Not Completed | 33 | 34 | 11 | 25
Not completed — Adverse Event | 5 | 6 | 0 | 0
Not completed — Extra exclusion criterion amended | 2 | 1 | 1 | 1
Not completed — Informed consent has been withdrawn | 2 | 2 | 1 | 1
Not completed — Patient is not able to attend visits | 8 | 9 | 7 | 6
Not completed — Patient´s compliance | 4 | 3 | 1 | 2
Not completed — Lost to Follow-up | 5 | 5 | 0 | 6
Not completed — PCR positive at week 24 | 0 | 0 | 0 | 1
Not completed — Other reason | 7 | 8 | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon/Ribavirin 800 mg (24 Weeks): Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 800 mg orally daily for 24 W. The untreated Follow-up was for 24 W.
- Total: Total of all reporting groups
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks) | Total
Number analyzed (Participants) | 151 | 144 | 33 | 52 | 380
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (11.1) | 35.7 (10.2) | 35.8 (11.2) | 35.2 (10.0) | 36.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 54 | 14 | 21 | 151
  Male | 89 | 90 | 19 | 31 | 229

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Sustained Virologic Response Rate At 24 Weeks Post Completion of the Treatment
Description: Sustained virological response was defined as the percentage of participants in each group with undetectable Hepatitis C virus-Ribonucleic acid (HCV-RNA) measurement at 24 weeks post completion of the treatment.
Time Frame: Up to Week 48 (24 weeks post completion of the treatment)
Population: Standard analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Percentage of participants | 80.9 [72.5 to 87.6] | 78.2 [69.3 to 85.5] | 81.0 [58.1 to 94.6] | 61.5 [40.6 to 79.8]
Statistical Analysis 1: Comparison: Peginterferon/Ribavirin 800 mg (16 Weeks) vs Peginterferon/Ribavirin 400 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — The statistical analysis was applied to Arms Peginterferon/Ribavirin 800 mg (16 weeks) and Peginterferon/Ribavirin 400 mg (16 weeks); Risk Difference (RD) = 32.0, 95% CI 2-sided [10.5 to 53.5]
Statistical Analysis 2: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (24 Weeks); Test type: Non-Inferiority or Equivalence — The statistical analysis was applied to arms Peginterferon/Ribavirin 800 mg (24 weeks) and Peginterferon/Ribavirin 400 mg (24 weeks); Risk Difference (RD) = -3.2, 95% CI 2-sided [-14.0 to 7.6]
Statistical Analysis 3: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 800 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — The statistical analysis was applied to arms Peginterferon/Ribavirin 800 mg (24 weeks) and Peginterferon/Ribavirin 800 mg (16 weeks); Risk Difference (RD) = 7.2, 95% CI 2-sided [-4.7 to 19.1]
Statistical Analysis 4: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — The statistical analysis was applied to arms Peginterferon/Ribavirin 800 mg (24 weeks) and Peginterferon/Ribavirin 400 mg (16 weeks); Risk Difference (RD) = -21.1, 95% CI 2-sided [-42.2 to -0.1]

2. Primary Outcome: Percentage of Participants With Hepatitis C Virus-RNA Determined by AMPLICOR HCV Test At Week 24 and Week 48
Description: Serum Hepatitis C Virus-RNA (HCV-RNA) was done by Polymerase chain reaction (PCR). Samples for a qualitative PCR (AMPLICOR® HCV Test v2.0) were obtained at Week 24 and Week 48. 'G2' and 'G3' indicates Genotype 2 and Genotype 3 respectively.
Time Frame: At Week 24 and Week 48
Population: Standard analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Percentage of participants
  G2, W24, HCV-RNA Positive (n=14,13,3,3) | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  G2, W24, HCV-RNA Negative (n=14,13,3,3) | 92.9 [66.1 to 99.8] | 100 [75.3 to 100] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  G2, W48, HCV-RNA Positive (n=14,13,3,3) | 7.1 [0.2 to 33.9] | 23.1 [5.0 to 53.8] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6]
  G2, W48, HCV-RNA Negative (n=14,13,3,3) | 92.9 [66.1 to 99.8] | 76.9 [46.2 to 95.0] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2]
  G3, W24, HCV-RNA Positive (n=101,97,18,23) | 1.0 [0.0 to 5.4] | 3.1 [0.6 to 8.8] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  G3, W24, HCV-RNA Negative (n=101,97,18,23) | 99.0 [94.6 to 100] | 96.9 [91.2 to 99.4] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  G3, W48, HCV-RNA Positive (n=101,97,18,23) | 20.8 [13.4 to 30.0] | 21.6 [13.9 to 31.2] | 11.1 [1.4 to 34.7] | 39.1 [19.7 to 61.5]
  G3, W48, HCV-RNA Negative (n=101,97,18,23) | 79.2 [70.0 to 86.6] | 78.4 [68.8 to 86.1] | 88.9 [65.3 to 98.6] | 60.9 [38.5 to 80.3]

3. Secondary Outcome: Percentage of Participants With Virological Response at the End of the Treatment
Description: Virological response at the end of the treatment (ETR) was defined as the percentage of participants with negative qualitative PCR in each group at completion of the treatment. ETR is defined as Week 16 and Week 24.
Time Frame: At Week 16 and Week 24
Population: Standard analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Percentage of participants | 98.3 [93.9 to 99.8] | 97.3 [92.2 to 99.4] | 95.2 [76.2 to 99.9] | 100 [86.8 to 100]
Statistical Analysis 1: Comparison: Peginterferon/Ribavirin 800 mg (16 Weeks) vs Peginterferon/Ribavirin 400 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 2: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (24 Weeks); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Risk Difference (RD) = -2.6, 95% CI 2-sided [-6.4 to 1.3]
Statistical Analysis 3: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 800 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.4 to 1.4]
Statistical Analysis 4: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (16 Weeks); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; Risk Difference (RD) = 0.6, 95% CI 2-sided [-0.5 to 1.7]

4. Secondary Outcome: Percentage of Participants With Virologic Response Rates as Per Genotype at End of Treatment
Description: Virologic Response was defined as undetectable HCV-RNA levels (determined by AMPLICOR HCV test) at Week 16 and Week 24. Virologic response rates based on genotype (G2 and G3) were reported. ETR is defined as Week 16 and Week 24.
Time Frame: At Week 16 and Week 24
Population: Standard analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Percentage of participants
  G2, W16, Virologic Response (n=14,13,3,3) | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 66.7 [9.4 to 99.2] | 100 [29.2 to 100]
  G2, W24, Virologic Response (n=14,13,3,3) | 92.9 [66.1 to 99.8] | 100 [75.3 to 100] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  G3, W16,Virologic Response (n=101,97,18,23) | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 100 [81.5 to 100] | 100 [85.2 to 100]
  G3, W24,Virologic Response (n=101,97,18,23) | 99.0 [94.6 to 100] | 96.9 [91.2 to 99.4] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

5. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 48
Population: The Safety analysis population was defined to include only participants who received at least one dose of (either) study medication and had at least one post-baseline assessment.
Measure: Number; unit: Number of Participants
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 144 | 141 | 30 | 48
Number of Participants
  Any AE | 139 | 138 | 29 | 45
  Any SAE | 12 | 18 | 0 | 2

6. Secondary Outcome: Median Hemoglobin Levels at End of Treatment
Description: Hemoglobin (Hb) levels at end of treatment (Week 16 and Week 24) were reported. The mean lowest Hb value after treatment starts with a median of 129 gram (g)/Litre (L). The far most frequent hemoglobin class was >=100 g/L. The purpose of assessing the Hb levels is associated with ribavirin dose. The primary toxicity of ribavirin dose (1000-1200 mg/day, maximum tolerated dose) is anemia with a reduction in hemoglobin levels generally occurring within the first 1-2 weeks of initiating therapy. Decreases in hemoglobin seen in the combination treatment of ribavirin and Interferon-alfa are managed with reduction in ribavirin dosage to 600 mg/day.
Time Frame: At Week 16 and Week 24
Population: The Safety analysis population was defined to include only participant who received at least one dose of (either) study medication and had at least one post-baseline safety assessment.
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 144 | 141 | 30 | 48
g/L
  At Week 16 | 123.00 [116.00 to 134.00] | 131.00 [120.50 to 140.00] | 129.50 [116.00 to 140.50] | 131.00 [124.00 to 143.00]
  At Week 24 | 124.00 [115.00 to 133.00] | 130.00 [121.00 to 140.00] | NA [NA to NA] — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA [NA to NA] — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.

7. Secondary Outcome: Mean SF-36 Scores at Baseline and Weeks 16, 24 and 48
Description: Short-Form Health Survey (SF-36) is a 36-item questionnaire measuring eight domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Where Baseline (BS) is Week 0.
Time Frame: At Baseline (Week 0) and Weeks 16, 24 and 48
Population: Standard analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Score on a scale
  G2, BS, Physical Functioning (n=14,13,3,3) | 87.8 (22.1) | 87.9 (12.9) | 76.7 (10.4) | 69.4 (43.2)
  G2, W16, Physical Functioning (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 63.3 (20.8) | 63.3 (31.8)
  G2, W24 Physical Functioning (n=14,13,3,3) | 73.5 (20.7) | 79.0 (17.9) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, Physical Functioning, (n=14,13,3,3) | 80.6 (30.3) | 81.0 (20.6) | 82.5 (17.7) | 85.0 (21.2)
  G3, BS, Physical Functioning (n=101,97,18,23) | 90.6 (13.9) | 85.9 (18.3) | 87.2 (15.2) | 77.9 (26.6)
  G3, W16, Physical Functioning (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 81.1 (14.5) | 69.8 (28.1)
  G3, W24, Physical Functioning (n=101,97,18,23) | 79.6 (20.8) | 79.8 (22.5) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3, W48, Physical Functioning (n=101,97,18,23) | 91.6 (13.8) | 89.7 (18.6) | 88.9 (12.9) | 87.9 (12.8)
  G2, BS,Role Functioning Physical (n=14,13,3,3) | 72.2 (38.4) | 88.9 (22.0) | 75.0 (25.0) | 50.0 (70.7)
  G2,W16,Role Functioning Physical (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 16.7 (28.9) | 41.7 (52.0)
  G2,W24,Role Functioning Physical (n=14,13,3,3) | 57.5 (31.3) | 50.0 (37.3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48,Role Functioning Physical (n=14,13,3,3) | 56.3 (47.7) | 88.9 (18.2) | 87.5 (17.7) | 87.5 (17.7)
  G3, BS,Role Functioning Physical (n=101,97,18,23) | 81.2 (30.7) | 73.9 (33.0) | 83.3 (28.0) | 75.0 (34.3)
  G3,W16,Role Functioning Physical (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 61.1 (35.6) | 61.8 (40.6)
  G3,W24,Role Functioning Physical (n=101,97,18,23) | 60.4 (40.4) | 63.6 (39.5) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3,W48,Role Functioning Physical (n=101,97,18,23) | 90.5 (23.9) | 85.5 (30.2) | 91.7 (17.7) | 81.3 (31.0)
  G2, BS, Bodily Pain (n=14,13,3,3) | 78.6 (29.0) | 83.0 (24.5) | 71.0 (25.7) | 61.0 (55.2)
  G2,W16, Bodily Pain (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 61.3 (39.0) | 54.3 (40.7)
  G2, W24, Bodily Pain (n=14,13,3,3) | 74.0 (28.5) | 55.5 (33.3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2, W48, Bodily Pain (n=14,13,3,3) | 76.1 (33.7) | 84.0 (15.6) | 81.0 (26.9) | 81.0 (26.9)
  G3, BS, Bodily Pain (n=101,97,18,23) | 85.5 (22.0) | 82.9 (19.7) | 73.0 (26.1) | 83.6 (30.6)
  G3, W16, Bodily Pain (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 69.6 (19.4) | 70.2 (31.6)
  G3, W24, Bodily Pain(n=101,97,18,23) | 76.7 (27.3) | 71.5 (25.9) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3,W48, Bodily Pain (n=101,97,18,23) | 89.5 (19.2) | 87.7 (23.0) | 84.1 (18.1) | 81.9 (33.3)
  G2,BS, General Health (n=14,13,3,3) | 60.4 (9.3) | 66.3 (17.6) | 62.3 (21.1) | 51.0 (36.8)
  G2,W16,General Health (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 42.3 (27.5) | 49.0 (21.3)
  G2, W24, General Health (n=14,13,3,3) | 63.2 (12.7) | 67.2 (20.5) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, General Health (n=14,13,3,3) | 76.3 (13.4) | 76.0 (14.9) | 53.5 (26.2) | 43.5 (26.2)
  G3, BS, General Health (n=101,97,18,23) | 67.2 (18.5) | 61.7 (19.4) | 56.9 (12.9) | 61.1 (23.6)
  G3, W16, General Health (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 58.3 (20.4) | 63.6 (19.9)
  G3, W24, General Health (n=101,97,18,23) | 68.1 (18.1) | 59.5 (21.3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3, W48, General Health (n=101,97,18,23) | 73.9 (16.0) | 70.5 (21.6) | 70.2 (19.5) | 63.0 (26.0)
  G2, BS, Vitality (n=14,13,3,3) | 58.1 (20.5) | 62.2 (11.4) | 43.3 (18.9) | 35.0 (49.5)
  G2,W16, Vitality (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 25.0 (21.8) | 30.6 (14.2)
  G2, W24, Vitality (n=14,13,3,3) | 38.5 (23.0) | 39.5 (22.0) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, Vitality (n=14,13,3,3) | 58.1 (19.3) | 63.9 (15.0) | 57.5 (24.7) | 45.0 (35.4)
  G3,BS, Vitality (n=101,97,18,23) | 55.8 (21.1) | 51.9 (21.4) | 51.7 (24.9) | 49.4 (24.8)
  G3,W16, Vitality (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 46.1 (19.5) | 43.5 (18.1)
  G3,W24, Vitality (n=101,97,18,23) | 46.9 (24.4) | 45.5 (23.8) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3, W48, Vitality (n=101,97,18,23) | 63.4 (19.1) | 58.7 (20.2) | 70.6 (15.7) | 60.1 (18.9)
  G2, BS, Social Functioning (n=14,13,3,3) | 80.6 (21.8) | 93.8 (10.6) | 75.0 (12.5) | 56.3 (44.2)
  G2, W16, Social Functioning (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 50.0 (43.3) | 58.3 (26.0)
  G2,W24, Social Functioning (n=14,13,3,3) | 63.8 (32.0) | 76.3 (28.5) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, Social Functioning (n=14,13,3,3) | 89.1 (15.6) | 86.1 (15.9) | 81.3 (26.5) | 81.3 (26.5)
  G3,BS, Social Functioning (n=101,97,18,23) | 83.8 (19.5) | 77.2 (23.5) | 86.1 (20.2) | 84.7 (20.8)
  G3, W16, Social Functioning (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 63.9 (20.2) | 66.9 (30.3)
  G3,W24, Social Functioning (n=101,97,18,23) | 68.8 (26.7) | 72.1 (26.3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3, W48, Social Functioning (n=101,97,18,23) | 86.6 (21.0) | 81.6 (27.0) | 87.5 (18.8) | 78.7 (26.8)
  G2, BS, Role Functioning Emotional (n=14,13,3,3) | 74.1 (36.4) | 88.9 (23.6) | 77.8 (19.2) | 50.0 (70.7)
  G2,W16, Role Functioning Emotional (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 33.3 (33.3) | 44.4 (50.9)
  G2,W24, Role Functioning Emotional (n=14,13,3,3) | 56.7 (38.7) | 43.3 (38.7) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, Role Functioning Emotional (n=14,13,3,3) | 60.4 (37.7) | 85.2 (24.2) | 100.0 (0.0) | 83.3 (23.6)
  G3,BS,Role Functioning Emotional (n=101,97,18,23) | 83.1 (29.7) | 73.2 (36.1) | 70.4 (35.1) | 68.5 (40.4)
  G3,W16,Role Functioning Emotional (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 63.0 (35.1) | 60.8 (41.2)
  G3,W24,Role Functioning Emotional (n=101,97,18,23) | 61.0 (41.0) | 57.4 (44.6) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3,W48,Role Functioning Emotional (n=101,97,18,23) | 90.9 (23.8) | 84.2 (33.4) | 88.9 (23.6) | 79.2 (36.3)
  G2,BS, Mental Health (n=14,13,3,3) | 66.5 (13.5) | 73.2 (14.9) | 57.3 (18.0) | 58.0 (48.1)
  G2,W16, Mental Health (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 42.7 (20.1) | 49.3 (19.7)
  G2,W24, Mental Health (n=14,13,3,3) | 59.2 (22.5) | 64.8 (21.2) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48, Mental Health (n=14,13,3,3) | 66.3 (19.2) | 76.1 (14.3) | 58.5 (37.5) | 70.0 (31.1)
  G3,BS, Mental Health (n=101,97,18,23) | 69.2 (16.6) | 67.8 (17.2) | 63.6 (17.4) | 59.6 (25.4)
  G3,W16, Mental Health (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 56.4 (15.0) | 55.5 (19.7)
  G3,W24, Mental Health (n=101,97,18,23) | 63.0 (19.9) | 63.2 (21.0) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3, W48, Mental Health (n=101,97,18,23) | 70.5 (15.7) | 68.8 (20.9) | 68.0 (20.2) | 64.1 (19.7)
  G2,BS,Reported Health Transition (n=14,13,3,3) | 2.7 (0.5) | 3.0 (0.8) | 3.7 (0.6) | 3.0 (2.8)
  G2,W16,Reported Health Transition (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 4.0 (1.0) | 3.0 (1.0)
  G2,W24,Reported Health Transition (n=14,13,3,3) | 2.6 (1.0) | 3.7 (0.8) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G2,W48,Reported Health Transition (n=14,13,3,3) | 1.8 (0.9) | 1.9 (0.8) | 2.0 (0.0) | 2.5 (0.7)
  G3,BS,Reported Health Transition (n=101,97,18,23) | 2.8 (1.1) | 2.9 (1.0) | 2.9 (0.9) | 2.8 (1.1)
  G3,W16,Reported Health Transition (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | 3.3 (1.1) | 2.9 (1.5)
  G3,W24,Reported Health Transition (n=101,97,18,23) | 3.0 (1.3) | 2.7 (1.4) | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a SF36 assessment for this group.
  G3,W48,Reported Health Transition (n=101,97,18,23) | 1.7 (0.9) | 1.9 (1.1) | 2.3 (1.2) | 2.2 (0.9)

8. Secondary Outcome: Mean FSS Scores at Baseline and Weeks 16, 24 and 48
Description: The Fatigue Severity Scale (FSS) is a self-administered instrument that includes 9 items rated on a 7-point scale, measuring fatigue severity. The participants were asked to score each statement, based on how the statement applied to them over the preceding week. The fatigue severity score is the average of the scores on the 9 questions; scores range from 1-7, with lower scores indicating less fatigue. Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0) and Weeks 16, 24 and 48
Population: Standard analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Score on a scale
  G2, BS (n=14,13,3,3) | 3.5 (1.2) | 3.4 (1.1) | 4.9 (0.3) | 3.9 (2.9)
  G2, W16 (n=14,13,3,3) | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | 6.2 (0.5) | 3.7 (1.8)
  G2, W24 (n=14,13,3,3) | 4.4 (1.3) | 4.4 (1.2) | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group.
  G2, W48 (n=14,13,3,3) | 3.4 (1.6) | 3.5 (1.2) | 4.5 (0.4) | 3.2 (2.8)
  G3,BS(n=101,97,18,23) | 3.6 (1.2) | 3.8 (1.6) | 3.4 (1.5) | 3.5 (1.6)
  G3, W16, (n=101,97,18,23) | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | 4.0 (1.6) | 4.3 (1.5)
  G3, W24 (n=101,97,18,23) | 4.1 (1.7) | 4.1 (1.7) | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group. | NA (NA) — The Protocol (and therefore the SAP) had not planned a FSS assessment for this group.
  G3, W48 (n=101,97,18,23) | 3.0 (1.3) | 3.2 (1.6) | 2.4 (1.6) | 3.7 (1.8)

9. Secondary Outcome: Mean Beschwerdeliste Score for Participants Receiving an Opioid Maintenance Therapy At Baseline and Weeks 16, 24 and 48
Description: Psychiatric assessment were performed using Beschwerdeliste (BL) questionnaires. BL results were analyzed descriptively by visit, treatment group, genotype and opioid maintenance therapy status. The BL questionnaire items were scored by calculating the average response to all answered items. Items were graded 1="stark" (affliction is strong) to 4="gar nicht" (not present). The higher the BL score, the less afflictions were present for a participant. Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0) and Weeks 16, 24 and 48
Population: Standard analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Score on a scale
  G2 ,BL, BS (n=14,13,3,3) | 3.3 (0.4) | 3.4 (0.5) | 3.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2, BL,W4 (n=14,13,3,3) | 3.1 (0.7) | 3.3 (0.4) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | 3.8 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2, BL, W8 (n=14,13,3,3) | 3.4 (0.7) | 3.6 (0.5) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2, BL, W12 (n=14,13,3,3) | 3.5 (0.7) | 3.3 (0.5) | 3.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2, BL,W24 (n=14,13,3,3) | 2.9 (0.6) | 3.2 (0.4) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2, BL,W48 (n=14,13,3,3) | 3.4 (0.4) | 3.4 (0.4) | 3.2 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | 4.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3, BL,BS(n=101,97,18,23) | 3.3 (0.4) | 3.3 (0.4) | 3.2 (0.2) | 3.3 (0.4)
  G3, BL,W4 (n=101,97,18,23) | 3.4 (0.6) | 3.0 (0.4) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3, BL,W8 (n=101,97,18,23) | 3.3 (0.6) | 3.0 (0.5) | 2.6 (0.3) | 3.7 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3, BL,W12 (n=101,97,18,23) | 3.2 (0.6) | 3.1 (0.5) | 3.2 (0.3) | 3.0 (0.5)
  G3,BL,W24 (n=101,97,18,23) | 3.2 (0.5) | 3.2 (0.5) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3,BL,W48 (n=101,97,18,23) | 3.6 (0.4) | 3.5 (0.4) | 3.4 (0.5) | 3.3 (0.5)

10. Secondary Outcome: Beck Depression Inventory Mean Score for Participants Receiving an Opioid Maintenance Therapy At Baseline and Weeks 4, 8, 12, 24 and 48
Description: For the psychiatric assessment, the results of the Beck Depression Inventory (BDI) questionnaires were evaluated. BDI results were analyzed descriptively by visit, treatment group, genotype and opioid maintenance therapy status. BDI is 21 item participant rated inventory evaluates depression symptoms, cognition, and physical symptoms of fatigue, weight loss, lack of interest in sex. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe. Total score: 0 to 63; higher score indicates more depression. Mean scores are presented by visit. Baseline is defined as Week 0.
Time Frame: At Baseline (Week 0) and Weeks 4, 8, 12, 24 and 48
Population: Standard analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 115 | 110 | 21 | 26
Score on a scale
  G2,BDI,BS (n=14,13,3,3) | 8.2 (4.0) | 5.4 (6.4) | 9.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2,BDI,W4 (n=14,13,3,3) | 10.7 (12.5) | 8.8 (9.7) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | 3.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2,BDI,W8 (n=14,13,3,3) | 10.0 (9.9) | 3.0 (4.2) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2,BDI,W12 (n=14,13,3,3) | 8.0 (9.9) | 8.5 (7.8) | 8.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2,BDI,W24 (n=14,13,3,3) | 11.5 (9.4) | 7.6 (4.7) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G2,BDI,W48 (n=14,13,3,3) | 3.8 (2.3) | 4.0 (5.1) | 4.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | 1.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3,BDI,BS (n=101,97,18,23) | 7.1 (6.4) | 8.9 (7.7) | 8.0 (5.5) | 7.0 (3.7)
  G3,BDI,W4 (n=101,97,18,23) | 7.9 (8.4) | 10.8 (8.1) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3,BDI,W8 (n=101,97,18,23) | 8.2 (8.5) | 12.7 (11.6) | 20.0 (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3,BDI,W12 (n=101,97,18,23) | 7.8 (7.3) | 11.4 (8.0) | 4.8 (5.3) | 15.0 (9.6)
  G3,BDI,W24 (n=101,97,18,23) | 8.0 (7.6) | 9.0 (7.9) | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group. | NA (NA) — Not Available. The Protocol (and therefore the SAP) had not planned an assessment for this group.
  G3,BDI,W48 (n=101,97,18,23) | 3.6 (4.7) | 6.7 (8.0) | 5.4 (7.7) | 6.6 (7.9)

11. Secondary Outcome: Time to Viral Response
Description: Time to viral response was calculated as Date of first negative PCR result after screening - date of PCR screening sample + 1 [in days]. Mean of number of days to viral response for overall population were reported.
Time Frame: Up to Week 48
Population: Standard analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Peginterferon/Ribavirin 800 mg (24 Weeks) | Peginterferon/Ribavirin 400 mg (24 Weeks) | Peginterferon/Ribavirin 800 mg (16 Weeks) | Peginterferon/Ribavirin 400 mg (16 Weeks)
Number analyzed (Participants) | 151 | 144 | 33 | 52
Days | 165.1 (73.6) | 165.0 (78.8) | 114.5 (76.7) | 122.8 (56.4)
Statistical Analysis 1: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (24 Weeks); Test type: Superiority or Other; p = 0.2667, Regression, Cox; Hazard Ratio (HR) = 0.6290
Statistical Analysis 2: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 800 mg (16 Weeks); Test type: Superiority or Other; p = 0.9999, Regression, Cox
Statistical Analysis 3: Comparison: Peginterferon/Ribavirin 800 mg (24 Weeks) vs Peginterferon/Ribavirin 400 mg (16 Weeks); Test type: Superiority or Other; p = 0.9891, Regression, Cox

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: An adverse event was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Groups:
- Ribavirin 800 mg/24W: Eligible participants were administered peginterferon alfa-2a (PEG-IFNα-2a) 180 microgram (mcg) subcutaneously (SC) once weekly + Ribavirin 800 milligram (mg) orally daily for 24 weeks (W). The untreated Follow-up was for 24 W.
- Ribavirin 400 mg/24W: Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 400 mg orally daily for 24 W. The untreated Follow-up was for 24 W.
- Ribavirin 800 mg/16W: Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 800 mg orally daily for 16 W. The untreated Follow-up was for 24 W.
- Ribavirin 400 mg/16W: Eligible participants were administered PEG-IFNα-2a 180 mcg SC once weekly + Ribavirin 400 mg orally daily for 16 W. The untreated Follow-up was for 24 W.
Arm/Group | Ribavirin 800 mg/24W | Ribavirin 400 mg/24W | Ribavirin 800 mg/16W | Ribavirin 400 mg/16W
Serious Adverse Events (participants affected / at risk) | 12/144 | 18/141 | 0/30 | 2/48
Other Adverse Events (participants affected / at risk) | 133/144 | 128/141 | 27/30 | 38/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin 800 mg/24W (N=144) | Ribavirin 400 mg/24W (N=141) | Ribavirin 800 mg/16W (N=30) | Ribavirin 400 mg/16W (N=48)
Perianal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis of arm (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pilonidal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative infection (Infections and infestations) | 1 | 0 | 0 | 0
Right otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Salmonella infection nos (Infections and infestations) | 1 | 0 | 0 | 0
Septic phlebitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcus aureus septicemia (Infections and infestations) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Epileptic seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure cerebral (Nervous system disorders) | 0 | 1 | 0 | 0
Tia (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain nos (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0
Acute and transient psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Dependence on opiates (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Lymphadenopathy hilar (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Renal anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Coronary disease (Cardiac disorders) | 1 | 0 | 0 | 0
Darier's disease (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Sudden deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Anterior cruciate ligament tear (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Opiate toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pregnancy of partner (Social circumstances) | 0 | 1 | 0 | 0
Breast cosmetic surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin 800 mg/24W (N=144) | Ribavirin 400 mg/24W (N=141) | Ribavirin 800 mg/16W (N=30) | Ribavirin 400 mg/16W (N=48)
Fatigue (General disorders) | 50 | 53 | 11 | 15
Flu like symptoms (General disorders) | 54 | 54 | 6 | 8
Fever (General disorders) | 17 | 13 | 8 | 9
Flu-like symptoms (General disorders) | 10 | 14 | 0 | 4
Injection site reaction (General disorders) | 5 | 7 | 0 | 0
Tiredness (General disorders) | 7 | 4 | 0 | 0
Depression (Psychiatric disorders) | 26 | 24 | 3 | 6
Sleep disorder (Psychiatric disorders) | 13 | 10 | 3 | 6
Insomnia (Psychiatric disorders) | 18 | 8 | 2 | 3
Depressed mood (Psychiatric disorders) | 8 | 8 | 1 | 2
Hair loss (Skin and subcutaneous tissue disorders) | 20 | 20 | 2 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 15 | 0 | 2
Exanthema (Skin and subcutaneous tissue disorders) | 13 | 10 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 11 | 2 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3
Seborrheic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 15 | 4 | 2
Diarrhea (Gastrointestinal disorders) | 13 | 11 | 0 | 1
Heartburn (Gastrointestinal disorders) | 5 | 9 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 1 | 0
Common cold (Infections and infestations) | 13 | 9 | 2 | 2
Bronchitis (Infections and infestations) | 1 | 4 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 2 | 0
Cephalgia (Nervous system disorders) | 20 | 26 | 7 | 8
Appetite lost (Metabolism and nutrition disorders) | 20 | 17 | 2 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13 | 13 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 13 | 9 | 0 | 1
Leucopenia (Blood and lymphatic system disorders) | 6 | 5 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 8 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 9 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 2 | 2
Loss of weight (Investigations) | 7 | 5 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 10 | 9 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.